CLINICAL TRIAL: NCT06166524
Title: Pulsed-field Catheter Ablation as the First-line Treatment for Asymptomatic Non-paroxysmal Atrial Fibrillation
Brief Title: Pulsed-field Ablation for Patients With Asymptomatic Non-paroxysmal Atrial Fibrillation
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Regional Hospital Liberec (Other); Nemocnice AGEL Trinec-Podlesi a.s. (Other); Brno University Hospital (Other); University Hospital Ostrava (Other); VFN (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PF-A-SYMPTOMATIC
Record Dates: First submitted 2023-09-21; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-09

CONDITIONS: Atrial Fibrillation; Pulsed-field Ablation; Functional Exercise Testing
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early invasive strategy (Active Comparator): Patients will undergo early catheter ablation for atrial fibrillation using pulsed-field ablation energy
  Interventions: Procedure: Catheter ablation for atrial fibrillation using pulsed-field energy
- Conservative arm (Placebo Comparator): Patients will undergo cardioversion with antiarrhythmic drug treatment. In patients with atrial fibrillation reoccurrence, an optimalization of bradycardia medication will be done using smart watches heart rate monitoring
  Interventions: Procedure: Conservative arm

INTERVENTIONS:
Procedure: Catheter ablation for atrial fibrillation using pulsed-field energy — Patients will undergo pulmonary vein isolation using pulsed-field energy
  Arms: Early invasive strategy
Procedure: Conservative arm — Patients will undergo electrical cardioversion with consequent treatment with antiarrhythmic drugs
  Arms: Conservative arm

SUMMARY:
The goal of the study is to test the hypothesis whether the treatment of patients with asymptomatic non-paroxysmal AF based on catheter ablation will be superior than conservative approach consisting of electrical cardioversion with AADs treatment in terms of significant improvement of functional exercise capacity. Secondary hypothesis is that mild functional improvement would be present also by achieving optimum heart rate by means of the titration of beta-blocker dose.

Patients with non-paroxysmal asymptomatic AF will be enrolled and randomized to either early invasive strategy arm (EIS;, i.e. catheter ablation), or conservative arm (CS; ie. cardioversion followed by antiarrhythmic drug treatment. As baseline examinations, functional cardiopulmonary exercise testing (CPET), Holter, recording, and echocardiography will be done. After one month, the procedure (catheter ablation or cardioversion) will be performed. Outpatients visits are scheduled at 3, 6, 9 and 12 months after the randomization. At each visit, ECG Holter recording will be done. CPET will be repeated at M3 and M12 visits. In patients in the CS arm with AF recurrence, the dose of BB will be optimized using smart watches (the goal < 110/min on average, but to achieve 75% of predicted maximum heart rate). The endpoint will be the change in VO2 max between baseline and 12M CPET. Secondary endpoints will be AF burden, AF freedom, the change in the concentration of NT-proBNP, the change in the left atrial diameter and left ventricular ejection fraction, the proportion of patients with no improvement while in SR, and the improvement in the quality-of-life at 12 months.

DETAILED DESCRIPTION:
Background According to the current guidelines, catheter ablation (CA) for atrial fibrillation (AF) is recommended for rhythm control therapy in patients with paroxysmal or non-paroxysmal AF to improve symptoms of AF recurrences. In asymptomatic AF patients, CA is only recommended for patients with reduced ejection fraction to improve survival. Still, no randomized study has shown benefits from CA in asymptomatic AF patients without left ventricular dysfunction. In a subanalysis of large, randomized EAST-AFNET 4 trial, a prognostic benefit was seen also in asymptomatic AF patients; however, i) the most often antiarrhythmic measure in this study were antiarrhythmic drugs (AADs) and not CA, and ii) the study compared the early AF treatment vs usual treatment (and not CA vs conservative treatment). Moreover, due to an occurrence of regular focal or re-enterant atrial tachycardia after CA that is more difficult to control, the symptoms could even worsen after catheter ablation of asymptomatic patients. Therefore, due to the absence of evidence of clear benefit and possible complications, CA is not recommended as the first-line treatment for asymptomatic AF patients.

Treatment of these patients varies significantly among cardiologist; some are referred for electrical cardioversion with or without treatment with AADs, while others are treated using a rate-control strategy, and finely, some of them are referred directly for CA. The effect of CA on QoL differs among studies: some reported substantial, other studies reported minor or no improvement of QoL after successful CA. A few observational studies on catheter ablation in asymptomatic AF patients have described improved functional capacity (VO2 max) determined using functional cardiopulmonary exercise testing (CPET). For instance, Fiala et al. reported an improvement in VO2 max by 3.4+4.7 ml/kg/min in 171 patients with long-standing persistent AF after CA who maintained SR. Similar improvement was reported in the cohort of 32 patients with persistent AF after successful CA followed by SR maintenance by Mohanty et al. No improvement in VO2 max were reported in both reports in patients with failed ablation and persistent AF recurrence.

For rate control in patients with failed ablation, beta-blockers or verapamil were mainly used to achieve sufficient rate-control. Heart rate lowering is very effective in patients with tachycardia-induced cardiomyopathy, on the other hand, the inability to increase the heart rate during exercise could lead to insufficient cardiac output during maximum exercise. For instance, in the recently published study on patients with heart failure with preserved ejection fraction of which 1/3 had a history of AF, the withdrawal of BB was associated with significant improvement in VO2 max during CPET.

Due to an absence of randomized studies, ESC guidelines do not recommend CA as the first-line treatment of AF in this asymptomatic AF patients.

The advent of pulsed-field ablation (PFA provides safe, very fast, and efficacious pulmonary vein isolation (PVI) and additional left atrial ablation. The present study will compare CA to conservative treatment in asymptomatic, non-paroxysmal AF patients.

Our primary hypothesis is that the treatment approach based on early invasive strategy (catheter ablation) in patients presented with asymptomatic AF will be superior than conservative approach consisting of electrical cardioversion with AADs treatment in terms of significant improvement of functional exercise capacity.

Patients Patients with asymptomatic non-paroxysmal AF will be enrolled. The absence of symptoms will be confirmed by a quality-of-life questionnaire (AFEQT > 80 points for inclusion). Furthermore, NT-BNP will be checked at enrollment, and only patients with a concentration of NT-pro BNP less than 800 pg/mL can be enrolled.

During baseline examinations, 5-day ECG Holter recording and symptom-limited CPET (CPET-1) will be done. The aim of the first CPET (CPET-1) will be to assess baseline VO2 max, and the results of S1 will serve the baseline value for primary endpoint analysis. At the first visit, patients will be randomized to the group EIS (early invasive strategy) or CS (conservative strategy).

In 4 weeks after the enrollment ( +/- 1 week), the index procedure will be done. Patients in the EIS group will undergo CA of AF. CA will be done in analgosedation or general anesthesia using pulsed-field energy by means of pentaspline ablation catheter (Farawave, BSCI, USA) and corresponding pulsed-field energy generator (Farapulse, BSCI, USA). The goal will be to achieve pulmonary vein isolation (entrance and exit block), additional ablation lesions (posterior wall isolation, mitral isthmus) will be left on the discretion of treating physician. AADs (but not amiodarone) can be used in this patient cohort after CA until the end of blanking period.

Patients in the CS group will undergo electrical cardioversion as it is routinely done (short general anesthesia, biphasic shock of 360 J, max. 3 attempts). If not contraindicated, AADs (with an exception of amiodarone) will be used in all patients after electrical cardioversion.

Blanking period The first 3 months after the index procedure will serve as blanking period. During this period, the use of non-amiodarone AADs or electrical cardioversion is allowed in both groups, but not CA. AADs will be stopped in the EIS group at the end of the blanking period.

Further outpatient follow-up The outpatient follow-up controls will be done at 3, 6, 9 and 12 months after randomization. Each control consists of routine cardiology examination, ECG recording and 5-day Holter recording. At 3-month control, an optional CPET (CPET-2) can be done, but only in patients in SR from CS arm. The reason is a very high AF recurrence in the CS arm, and the purpose of CPET-2 is to assess the potential improvement in VO2max in the CS patients while in SR.

Any antiarrhythmic measure, i.e. re-initiation of antiarrhythmic drugs in the EIS arm, cardioversion or ablation for AF in both arms, could be done solely only if patients present with at least moderate symptoms clearly related to AF. In asymptomatic patients, rate-control strategy will be used, if AF reoccurs. In patients with AF reoccurrence in the CS arm, the optimal dose of beta-blockers (or other bradycardia medication) will be optimized using smart watches monitoring. All CS patients with AF reoccurrence will get smart watches for 2 months to daily monitor the heart rate at rest, at night, and during exercise. The purpose of this measure is to achieve the rest rate less than 110/min on average, but to enable the increase of heart rate up to 75% of maximum heart rate.

For the purpose to assess the maximum heart rate during exercise, data from the CPET-1 and the baseline Holter recording will be used.

Five-day ECG Holter monitoring will be done at 3, 6, 9 and 12 months. At the 12-month control, the last functional CPET (CPET-3) will be done. At the same control, echocardiography examination will be done, blood samples for NT-pro BNP analysis will be drawn, and all patients will be asked to fill the QoL questionnaire assessing changes in QoL during the study period.

The main goal is to compare the results of functional CPET between baseline (CPET-1) and 12 months (CPET-3) between groups.

Primary endpoints:

The change in VO2 max during functional CPET between baseline and 12-month examination (CPET-1 vs CPET-2) between both groups Secondary endpoints

1. the time to the first AF reoccurrence (AF reoccurrence is defined as AF lasing more than 30 sec on any Holter recording or during follow-up examination)
2. AF burden. AF burden is defined as percentage in time spent in AF during Holter recordings.
3. the proportion of really asymptomatic patients. It means patients without any improvement (either subjective or at CPET) during SR compared to baseline.
4. the difference in VO2 max between CPET-1 and CPET-3 in patients with AF reoccurrence, in whom BB optimization was done suing smart watches
5. the improvement in the quality of life assessed at 12-month examination between groups
6. the changes in the concentration of NT-proBNP between baseline and 12 months between groups
7. the changes in the left atrial dimension and left ventricular ejection fraction between baseline and 12 month examinations between groups

ELIGIBILITY:
Inclusion Criteria:

* non-paroxysmal AF
* absence of symptoms during standard clinical evaluation
* AFEQT> 80
* NT-pro BNP < 800 pg/mL

Exclusion Criteria:

* significant valvular disease
* left ventricular dysfunction - LV EF < 50 %
* history of tachycardia - induced cardiomyopathy
* pulmonary hypertension (sPAP > 40 mm Hg)
* age > 75 years
* LA size > 60 mm
* physical limitations that don't enable functional cardiopulmonary exercise testing
* overt coronary artery disease
* pregnancy
* BMI > 40
* chronic obstructive pulmonary disease with moderate or severe obstruction
* life expectancy less than 2 years
* permanent AF
* ophthalmological medication (eye drops) containing beta-blockers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in VO2 max | 12 months
  The change in VO2 max during baseline and 12 month functional CardioPulmonary Exercise Testing

SECONDARY OUTCOMES:
Sinus rhythm maintenance | 12 monthhs
  The time to the first reoccurrence of atrial fibrillation
AF burden | 12 months
  The percentage of time spent in atrial fibrillation during all Holter recordings
Proportion of really asymptomatic patients | 12 months
  The proportion of patients with no significant improvement during cardiopulmonary exercise testing while in SR, and no subjectively reported improvement
VO2 max change in patients with atrial fibrillation reoccurrence | 12 months
  Change in VO2 max between the cardiopulmonary exercise testing at baseline and at 12 months in patients, who had atrial fibrillation reoccurrence and in whom bradycardia medication was optimized
NT-pro BNP | 12 months
  Change in the concentrations of NT-pro BNP between baseline and 12 month examinations, comparison between groups
Left atrial dimension and left ventricular ejection fraction | 12 months
  Changes in the left atrial dimension and left ventricular ejection fraction between baseline and 12 examinations, comparison between groups

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Osmančík, Principal Investigator — Cardiac center University Hospital Kralovske Vinohrady
Locations (1):
- Cardiocenter, 3rd Medical School, Charles University and University Hospital Kralovske Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
The study data can be shared 6 months after the study completion
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data will be available six months after study publication

REFERENCES:
- [Result] Kirchhof P, Camm AJ, Goette A, Brandes A, Eckardt L, Elvan A, Fetsch T, van Gelder IC, Haase D, Haegeli LM, Hamann F, Heidbüchel H, Hindricks G, Kautzner J, Kuck KH, Mont L, Ng GA, Rekosz J, Schoen N, Schotten U, Suling A, Taggeselle J, Themistoclakis S, Vettorazzi E, Vardas P, Wegscheider K, Willems S, Crijns HJGM, Breithardt G; EAST-AFNET 4 Trial Investigators. Early Rhythm-Control Therapy in Patients with Atrial
- [Result] Fiala M, Bulkova V, Sknouril L, Nevralova R, Toman O, Januska J, Spinar J, Wichterle D. Functional improvement after successful catheter ablation for long-standing persistent atrial fibrillation. Europace. 2017 Nov 1;19(11):1781-1789. doi: 10.1093/europace/euw282. PMID 27707782
- [Result] Wokhlu A, Monahan KH, Hodge DO, Asirvatham SJ, Friedman PA, Munger TM, Bradley DJ, Bluhm CM, Haroldson JM, Packer DL. Long-term quality of life after ablation of atrial fibrillation the impact of recurrence, symptom relief, and placebo effect. J Am Coll Cardiol. 2010 May 25;55(21):2308-16. doi: 10.1016/j.jacc.2010.01.040. PMID 20488300